CLINICAL TRIAL: NCT02528890
Title: Group B Streptococcal Carrier State Prevalence Among Arab Pregnant Women in Northern Israel District
Acronym: GBS
Status: Completed | Type: Observational
Sponsor: The Nazareth Hospital, Israel (Other)
Responsible Party: Principal Investigator, Marwan Hakim, Dr., The Nazareth Hospital, Israel
Other Study IDs: 15-2015
Record Dates: First submitted 2015-08-07; First posted 2015-08-19 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Streptococcus B Carrier State Complicating Pregnancy
Keywords: group B streptococcus; GBS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- preganat women between 34 - 40 weeks: Eligible pregnant women, who meet the inclusion criteria, will have a vaginal/anal swab taken to identify positive GBS carriers by PCR (polymerase chain reaction) test.
  Interventions: Other: vaginal/anal swab for GBS from all participants

INTERVENTIONS:
Other: vaginal/anal swab for GBS from all participants — All eligible pregnant women, who meet the inclusion criteria and gave their informed consent to participate in the study has to complete a questionnaire and have a vaginal / anal swab taken to identify positive GBS carriers by PCR (polymerase chain reaction) test.

SUMMARY:
The incidence of early neonatal GBS (group B Streptococcus) infection in the Nazareth Hospital through the years 2006-2013 has been higher compared to the national average. On reviewing all the cases of infants with early GBS infection, revealed that some of these infants were born to mothers who are not included in any of the high-risk groups that need to have prophylactic antibiotic treatment before delivery. Therefore, the question was whether pregnant Arab women in the North district of Israel have a higher GBS carrier state rate than the general rate in Israel?

DETAILED DESCRIPTION:
Signs of early onset GBS infection of the newborn appear during the first week of life. Usually, the bacteria pass from a GBS carrier mother to the newborn during labor. The infection can cause multi-system problems such as pneumonia, meningitis and even death of the newborn. The prevention of the disease is best achieved by prophylactic antibiotics administered to the mother during labor.

In order to prevent early onset GBS infection of the newborn, pregnant women are treated with preventive antibiotics during labor based on either of two protocols:

A. Risk factors: Women with risk factors such as premature birth, prolonged premature rupture of membranes, intra-partum maternal fever or a previous child with GBS infection are treated.

B. Universal screening: Towards the end of pregnancy, at 35 - 37th week, a vaginal/anal swab for GBS is taken, and those found positive will be treated.

According to the Israeli Ministry of Health regulations' from July 2005 it is not accepted to routinely perform screening for GBS in pregnant women at 35-37th week of pregnancy. Therefore, the Israeli approach to prevent early neonatal GBS infection is based mainly on antibiotic prophylaxis treatment during labor of all pregnant women with risk factors.

In a study conducted at the Western Galilee Medical Center in the city of Nahariya and published in 2006, there was a significant increase in the GBS carrier state rate compared to previously published studies. It was also found that higher GBS carrier state rates prevail among Arab women compared to Jewish women.

The primary question of this study is to calculate GBS carrier state prevalence among pregnant Arab women attending the labor ward at the Nazareth Hospital at the 34 to 40th week of their pregnancy.

A vaginal / anal swab will be taken from all eligible participants to identify GBS carriers by PCR (polymerase chain reaction) test.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 40
2. Origin: Arab
3. Gestational age: 34 to 40

Exclusion Criteria:

1. Rupture of membranes
2. Women in active labor who has had one or more vaginal examinations.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will include 184 participants who meet the inclusion criteria and gave their informed consent to participate. The sample size enables a confidence level of 95% within a 5% range of the GBS carrier rate, assuming that the rate is close to 17%. The investigators assume to identify 23 to 41 carriers, which will allow comparison of demographic variables between carriers and non-carriers.
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
percentage of participants with positive GBS swab | one year
  GBS swab results are: "+" = positive, which means the participant is a carrier for GBS or "-" = negative, which means the participant is not a carrier for GBS

CONTACTS AND LOCATIONS:
Overall Officials: Marwan M Hakim, MD, DSc, Principal Investigator — Nazareth Hospital EMMS
Locations (1):
- Nazareth Hospital, Nazareth, Israel